CLINICAL TRIAL: NCT05731128
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled Parallel-group Study to Evaluate the Efficacy and Safety of Dupilumab Therapy in Patients With Moderately to Severely Active Ulcerative Colitis With an Eosinophilic Phenotype
Brief Title: A Study to Investigate the Efficacy and Safety of Dupilumab Therapy Compared With Placebo in Participants Aged ≥18 Years With Moderately to Severely Active Ulcerative Colitis With an Eosinophilic Phenotype (LIBERTY-UC SUCCEED (Study in UC for Clinical Efficacy Evaluation of Dupilumab))
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT17746; U1111-1278-4042 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-02-03; First posted 2023-02-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Colitis Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dupilumab (Experimental): Initial loading dose followed by regular administration for the duration of the treatment period.
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): Initial loading dose followed by regular administration for the duration of the treatment period.
  Interventions: Drug: Placebo
- Open-label arm (optional) (Other): Regular administration of open label dupilumab
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — injection solution subcutaneous
  Other Names: Dupixent
  Arms: Dupilumab; Open-label arm (optional)
Drug: Placebo — injection solution subcutaneous
  Arms: Placebo

SUMMARY:
The protocol of this Phase 2 clinical trial consists of a double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the efficacy and safety of dupilumab in participants with moderately to severely active Ulcerative Colitis (UC) with an eosinophilic phenotype.

Screening period: 2 to up to 4 weeks

Treatment period:

52-week investigational medicinal product (IMP) intervention (dupilumab or matching placebo) from Week 0 to Week 52 Open-label arm (optional): administration of open-label dupilumab therapy for study participants who qualify. Follow-up period: 12 weeks The maximum duration of study per participant is up to 68 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥18 years of age at the time of signing the informed consent.
* Evidence of biomarker enrichment at time of screening.
* Moderately to severely active UC, defined as a baseline modified Mayo score of 5 to 9, inclusive, using the Mayo endoscopic subscore assigned during the concurrent local and central reading of the video endoscopy.
* Has a screening endoscopy with ≥2 endoscopic subscore in the Mayo score component assessment as determined by concurrent local and central reading of the video endoscopy.
* Has a baseline rectal bleeding subscore of ≥1 and baseline a stool frequency score of ≥1 as determined by the Mayo score component assessment.
* Participants with inadequate response/non-response, loss of response, or are intolerant of standard biologic therapy for their UC AND/OR Inadequate or non-responders, have shown loss of response, or are intolerant to at least 1 of the following treatments: oral corticosteroids (≤20 mg/day), 5-aminosalicylic acid (ASA) compounds, immunomodulators, small molecules.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Severe extensive colitis as evidenced by:

  * Current hospitalization
  * Likely to require surgery for the treatment of UC within 12 weeks of Screening Visit
* UC limited to the rectum only or to <20 cm of the colon as determined by central reading.
* Presence of an ileal pouch, ostomy, stoma or fistula or history of a fistula.
* Require, or required within the 2 months before screening, surgery for active gastrointestinal bleeding, peritonitis, intestinal obstruction, or intra-abdominal or pancreatic abscess requiring surgical drainage, or other conditions possibly confounding the evaluation of benefit from study agent treatment.
* Has a prior medical history of eosinophilic colitis.
* Participants with abdominal abscess, fulminant disease, or toxic megacolon.
* Participants with intestinal failure or short bowel syndrome.
* Presence of symptomatic colonic or small bowel obstruction, confirmed by objective radiographic or endoscopic evidence of a stricture with resulting obstruction (dilation of the colon or small bowel proximal to the stricture on barium radiograph or an inability to traverse the stricture at endoscopy).
* History of extensive colonic resection (eg, less than 30 cm of colon remaining) that would prevent adequate evaluation of the effect of study agent on clinical disease activity.
* History of colonic mucosal dysplasia or presence of adenomatous colonic polyps not removed OR presence of colonic mucosal dysplasia or adenomatous colonic polyps not removed during colonoscopy at screening visit.
* If the participant has extensive colitis for ≥8 years or disease limited to left side of colon (ie, distal to splenic flexure) for >10 years, regardless of age, a colonoscopy within 1 year of the screening visit is required to survey for dysplasia. Participants with dysplasia or cancer identified on biopsies will be excluded.
* Diagnosis of indeterminate colitis, microscopic colitis, ischemic colitis, or Crohn's disease or clinical findings suggestive of Crohn's disease.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-02-19 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving clinical response at Week 24 | Week 24
  Clinical response by modified Mayo score is defined as a decrease from baseline in the modified Mayo score of ≥2 points and at least a 30% reduction from baseline, and a decrease in rectal bleeding subscore of ≥1 OR an absolute rectal bleeding subscore of 0 or 1. The modified Mayo score consists of 3 subscores; a patient-reported subscore for rectal bleeding, a patient-reported subscore for stool frequency, and a Mayo endoscopic subscore. Each subscore ranges 0-3 with higher scores indicating greater disease severity. The total modified Mayo score ranges 0-9 with higher scores indicating greater disease severity.

SECONDARY OUTCOMES:
Proportion of participants who are in clinical response at Week 52 | Week 52
  Clinical response by modified Mayo score is defined as a decrease from baseline in the modified Mayo score of ≥2 points and at least a 30% reduction from baseline, and a decrease in rectal bleeding subscore of ≥1 OR an absolute rectal bleeding subscore of 0 or 1. The modified Mayo score consists of 3 subscores; a patient-reported subscore for rectal bleeding, a patient-reported subscore for stool frequency, and a Mayo endoscopic subscore. Each subscore ranges 0-3 with higher scores indicating greater disease severity. The total modified Mayo score ranges 0-9 with higher scores indicating greater disease severity.
Proportion of participants who are in clinical remission at Week 24 and Week 52 | Week 24 and Week 52
  Clinical remission by modified Mayo score is defined as a modified Mayo score of ≤2 with a stool frequency score ≤1, a rectal bleeding score = 0, AND a Mayo endoscopic subscore ≤1 with absence of friability. The modified Mayo score consists of 3 subscores; a patient-reported subscore for rectal bleeding, a patient-reported subscore for stool frequency, and a Mayo endoscopic subscore. Each subscore ranges 0-3 with higher scores indicating greater disease severity. The total modified Mayo score ranges 0-9 with higher scores indicating greater disease severity.
Proportion of participants in symptomatic remission over time | Baseline up to Week 52
  Symptomatic remission is defined as Mayo stool frequency score = 0, or Mayo stool frequency score = 1 with a ≥1-point decrease from baseline, and Mayo rectal bleeding score = 0.
Proportion of participants achieving histologic-endoscopic healing at Week 24, and Week 52 | Week 24 and Week 52
  Histologic-endoscopic healing is defined by Mayo endoscopic subscore of 0 or 1 and histological healing (Geboes score <2). Mayo endoscopic subscore ranges 0-3 with higher scores indicating greater disease severity. The Geboes Index score is a six-grade classification system for inflammation: Grade 0 - structural change only; Grade 1 -chronic inflammation; Grade 2 - lamina propria neutrophils; Grade 3 - neutrophils in epithelium; Grade 4 - crypt destruction; and Grade 5 - erosions or ulcers.
Proportion of participants with a Mayo endoscopic subscore of 0 or 1 without friability at Week 24, and Week 52 | Week 24 and Week 52
  The Mayo endoscopic subscore ranges 0-3 with higher scores indicating greater disease severity.
Proportion of participants with a Mayo endoscopic subscore of 0 at Week 24, and Week 52 | Week 24 and Week 52
  The Mayo endoscopic subscore ranges 0-3 with higher scores indicating greater disease severity.
Change from baseline in the partial Mayo score at Week 8, Week 24, and Week 52 | Baseline to Week 8, Week 24 and Week 52
  The partial Mayo score consists of 3 subscores; a patient-reported subscore for rectal bleeding, a patient-reported subscore for stool frequency, and a Physician's global assessment (PGA) subscore. Each subscore ranges 0-3 with higher scores indicating greater disease severity. The partial Mayo score ranges 0-9 with higher scores indicating greater disease severity.
Proportion of participants in clinical remission at Week 52 who are off concomitant oral corticosteroids (OCS) at least 4 weeks prior to Week 52 | Baseline up to Week 52
  Clinical remission by modified Mayo score is defined as a modified Mayo score of ≤2 with a stool frequency score ≤1, a rectal bleeding score = 0, AND a Mayo endoscopic subscore ≤1 with absence of friability. The modified Mayo score consists of 3 subscores; a patient-reported subscore for rectal bleeding, a patient-reported subscore for stool frequency, and a Mayo endoscopic subscore. Each subscore ranges 0-3 with higher scores indicating greater disease severity. The total modified Mayo score ranges 0-9 with higher scores indicating greater disease severity.
Proportion of participants in clinical remission at Week 52 who are off concomitant oral corticosteroids (OCS) at least 4 weeks prior to Week 52 among participants receiving OCS at baseline | Baseline up to Week 52
  Clinical remission by modified Mayo score is defined as a modified Mayo score of ≤2 with a stool frequency score ≤1, a rectal bleeding score = 0, AND a Mayo endoscopic subscore ≤1 with absence of friability. The modified Mayo score consists of 3 subscores; a patient-reported subscore for rectal bleeding, a patient-reported subscore for stool frequency, and a Mayo endoscopic subscore. Each subscore ranges 0-3 with higher scores indicating greater disease severity. The total modified Mayo score ranges 0-9 with higher scores indicating greater disease severity.
Change from baseline in abdominal pain assessed by Abdominal Pain Numerical Rating Scale (NRS) at Week 8, Week 24, and Week 52 | Baseline to Week 8, Week 24 and Week 52
  Abdominal pain NRS is a single item patient report outcome (PRO) tool that patients will use to report intensity of their worst abdominal pain during a daily recall period with 0 being 'no pain' and 10 being the 'worst pain imaginable'.
Incidence of treatment-emergent adverse events (TEAEs) or serious adverse events (SAEs) | Baseline up to Week 64
Concentration of dupilumab in serum over time. | Baseline up to Week 64
Incidence of treatment-emergent antidrug antibodies (ADA) against dupilumab. | Baseline up to Week 64
Change from baseline (Screening visit) in the normalized enrichment scores (NES) in type 2 inflammation transcriptome signature at Week 24 and Week 52. | Baseline to Week 24 and Week 52
  NES is a summary score of the expression of a specified set of genes defining a molecular phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (77):
- United States (27):
  - Om Research- Site Number : 8400029, Apple Valley, California
  - TLC Clinical Research- Site Number : 8400020, Beverly Hills, California
  - Om Research - Oxnard- Site Number : 8400028, Oxnard, California
  - Palmtree Clinical Research- Site Number : 8400048, Palm Springs, California
  - Clinical Trials Management Services - Thousand Oaks- Site Number : 8400034, Thousand Oaks, California
  - Homestead Associates in Research- Site Number : 8400004, Homestead, Florida
  - Wellness Clinical Research - Miami Lakes - 8181 Northwest 154th Street- Site Number : 8400009, Miami Lakes, Florida
  - GI Pros- Site Number : 8400046, Naples, Florida
  - Advanced Research Institute - New Port Richey- Site Number : 8400026, New Port Richey, Florida
  - Digestive Disease Consultants - Orange Park- Site Number : 8400042, Orange Park, Florida
  - Tellabio International Research Services- Site Number : 8400041, Pembroke Pines, Florida
  - GCP Clinical Research- Site Number : 8400014, Tampa, Florida
  - Gastroenterology Consultants - Roswell- Site Number : 8400022, Roswell, Georgia
  - Sanmora Bespoke Clinical Research Solutions- Site Number : 8400043, East Orange, New Jersey
  - Smart Medical Research - New York- Site Number : 8400037, Jackson Heights, New York
  - DiGiovanna Family Care- Site Number : 8400006, Massapequa, New York
  - Tryon Medical Partners - Charlotte - Piedmont Row Drive South- Site Number : 8400008, Charlotte, North Carolina
  - Care Access - Lumberton- Site Number : 8400018, Lumberton, North Carolina
  - UPMC Presbyterian- Site Number : 8400038, Pittsburgh, Pennsylvania
  - Advanced Gastroenterology Associates - Decatur- Site Number : 8400047, Decatur, Texas
  - Katy Integrative Gastroenterology- Site Number : 8400027, Katy, Texas
  - Medrasa Clinical Research - Medrasa Sherman- Site Number : 8400039, Sherman, Texas
  - Texas Digestive Disease Consultants - Southlake- Site Number : 8400013, Southlake, Texas
  - Digestive Health Specialists of Tyler- Site Number : 8400031, Tyler, Texas
  - Victoria Gastroenterology- Site Number : 8400019, Victoria, Texas
  - Washington Gastroenterology - Bellevue- Site Number : 8400025, Bellevue, Washington
  - Washington Gastroenterology - Tacoma- Site Number : 8400030, Tacoma, Washington
- Argentina (6):
  - Investigational Site Number : 0320006, Mar del Plata, Buenos Aires
  - Investigational Site Number : 0320001, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320004, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320007, Buenos Aires
  - Investigational Site Number : 0320008, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
- Canada (4):
  - Investigational Site Number : 1240007, Edmonton, Alberta
  - Investigational Site Number : 1240010, Scarborough Village, Ontario
  - Investigational Site Number : 1240006, Montreal, Quebec
  - Investigational Site Number : 1240003, Montreal, Quebec
- Chile (5):
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Concepción, Región del Biobío
- Japan (10):
  - Investigational Site Number : 3920006, Nagoya, Aichi-ken
  - Investigational Site Number : 3920005, Kashiwa, Chiba
  - Investigational Site Number : 3920008, Kitakyushu, Fukuoka
  - Investigational Site Number : 3920002, Sapporo, Hokkaido
  - Investigational Site Number : 3920001, Sapporo, Hokkaido
  - Investigational Site Number : 3920011, Kamakura, Kanagawa
  - Investigational Site Number : 3920010, Shimizu, Shizuoka
  - Investigational Site Number : 3920004, Bunkyo, Tokyo
  - Investigational Site Number : 3920007, Kyoto
  - Investigational Site Number : 3920009, Saitama
- Mexico (5):
  - Investigational Site Number : 4840005, Saltillo, Coahuila
  - Investigational Site Number : 4840002, Torreón, Coahuila
  - Investigational Site Number : 4840007, Guadalajara, Jalisco
  - Investigational Site Number : 4840004, Mexico City, Mexico City
  - Investigational Site Number : 4840003, Chihuahua City
- University of Puerto Rico - Medical Sciences Campus- Site Number : 6300002, San Juan, Puerto Rico
- South Africa (9):
  - Investigational Site Number : 7100005, Cape Town
  - Investigational Site Number : 7100009, Cape Town
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100007, Cape Town
  - Investigational Site Number : 7100006, Johannesburg
  - Investigational Site Number : 7100001, Johannesburg
  - Investigational Site Number : 7100008, Kempton Park
  - Investigational Site Number : 7100003, Port Elizabeth
  - Investigational Site Number : 7100004, Pretoria
- South Korea (5):
  - Investigational Site Number : 4100003, Haeundae-gu, Busan
  - Investigational Site Number : 4100005, Daegu, Daegu
  - Investigational Site Number : 4100006, Daejeon, Daejeon
  - Investigational Site Number : 4100002, Wŏnju, Gangwon-do
  - Investigational Site Number : 4100004, Daegu, Gyeongsangbuk-do
- Investigational Site Number : 1580002, Taichung, Taiwan
- Turkey (Türkiye) (4):
  - Investigational Site Number : 7920003, Gaziantep
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920001, Mersin
  - Investigational Site Number : 7920006, Zonguldak

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT17746 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25215&tenant=MT_SNY_9011